CLINICAL TRIAL: NCT01416896
Title: New Needle for Two-Needle Hemodialysis
Acronym: BME-1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomedical Enterprises Inc (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Alfredo Zarate, MD, Biomedical Enterprises Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BME-1; R44DK059062 (NIH)
Record Dates: First submitted 2011-08-09; First posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: End Stage Renal Disease
Keywords: End stage Renal Disease; Hemodialysis; Oxidative Stress; Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New venous needle, the "BME needle" (Experimental): Hemodialysis using the new venous needle, the "BME needle".
  Interventions: Procedure: Hemodialysis using a new venous needle, the "BME needle"
- Standard venous needle, the "standard needle" (Active Comparator): One hemodialysis using the standard venous needle, the "standard needle" (device).
  Interventions: Procedure: Hemodialysis using the standard venous needle

INTERVENTIONS:
Procedure: Hemodialysis using the standard venous needle — Hemodialysis using the standard venous dialysis needle
  Other Names: hemodialysis using the standard venous dialysis needle
  Arms: Standard venous needle, the "standard needle"
Procedure: Hemodialysis using a new venous needle, the "BME needle" — Hemodialysis using a new venous dialysis needle or the "BME needle"
  Other Names: The "BME needle" is a newly designed venous dialysis needle.
  Arms: New venous needle, the "BME needle"
Procedure: Hemodialysis using a new venous needle, the "BME needle" — One hemodialysis using a new venous needle, the "BME needle"
  Arms: New venous needle, the "BME needle"
Procedure: Hemodialysis using the standard venous needle — One hemodialysis using the standard venous needle
  Arms: Standard venous needle, the "standard needle"

SUMMARY:
Our preliminary studies have demonstrated that an innovative new design of the hemodialysis venous needle (the needle that returns the cleaned blood from the hemodialysis filter to the patient) with three jets is superior to the standard venous needle because it decreases the velocity and turbulence of the blood when compared with the standard venous needle, it is more efficient in the removal of toxins from the blood, and it is safe and effective. More importantly, our preliminary studies suggested that the new needle causes less damage to the dialysis vascular access and to circulating blood cells and less inflammation and oxidative stress. These will decrease medical complications, the high cost of care and death in dialysis patients. The current study will corroborate the finding of previous studies.

ELIGIBILITY:
Inclusion Criteria:(1) end stage renal disease receiving hemodialysis in an ambulatory outpatient dialysis facility (2) male or female, (3) ages 18-80, (4) arterio-venous graft or AV fistula as vascular access,

Exclusion Criteria:patients with fever, infection, inflammation or malignancy will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Net change in intracellular oxidative stress and intracellular proinflammatory cytokines levels | 4 hours of hemodialysis
  The net change in the levels of intracellular IL-6, IL-6 soluble receptor, IL-6 gp130, superoxide, H2O2 and IL-1 during dialysis (difference between pre and post dialysis) using the new venous needle will be compared with the change using the current venous needle.

SECONDARY OUTCOMES:
Net change in oxidative stress and proinflammatory cytokines in plasma | 4 hours hemodialysis
  The net change in the plasma levels of IL-1, IL-6, MDA and AOPP during dialysis (difference between pre and post dialysis) using the new venous needle will be compared with the net change that occurs in patients using the current venous needle

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo R Zarate, MD, Principal Investigator — Biomedical Enterprises Inc; Pedro A Jose, MD, PhD, Principal Investigator — Children National Medical Center
Locations (1):
- DaVita K Street Dialysis Center, Washington D.C., District of Columbia, United States